# **Study Protocol**

Unique Protocol ID: STUDY20190922

# NCT05469438

Brief Title: IMAS Optimization and Applicability in Acute and Subacute Stroke.

Official Title: IMAS Optimization and Applicability in Acute and Subacute Stroke.

Document Date: January 2, 2019



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke | | |
|---|---|---|---|
| Approved: | 01/2019 | Prior Version: | 10/2018 |

[USE THIS BIOMEDICAL PROTOCOL TEMPLATE IF YOUR PROJECT INVOLVES ANY PHYSICAL CONTACT OR MEDICAL INTERVENTIONS WITH PARTICIPANTS]

#### INSTRUCTIONS:

- Depending on the nature of your research, some sections may not be applicable to your research. Mark these sections with, "N/A" or leave blank as indicated.
- When you write a protocol, keep an electronic copy. You will need to modify this copy when
  making changes.

#### PROTOCOL TITLE:

IMAS Optimization and Applicability in Acute and Subacute Stroke.

#### PRINCIPAL INVESTIGATOR:

Salim Hayek, M.D., Ph.D.
Department of Anesthesiology
University Hospitals Cleveland Medical Center Case Western Reserve University
11100 Euclid Ave
Cleveland, OH 44106
(216)844-3771, Salim.Hayek@UHhospitals.org

Ciro Ramos Estebanez, MD., Ph.D., MBA, FNCS. Department of Neurology and Rehabilitation University of Illinois Hospital 1740 W. Taylor St. Chicago, IL 60612 (312).355.1528 cramoses@uic.edu

# UH FACULTY ADVISOR:

If the principal investigator's primary role at UH is resident, fellow or student, identify a faculty advisor.

N/A

# OTHER DEPARTMENTS INVOLVED IN THIS STUDY (IF APPLICABLE):

Department of Neurology (Cleveland VA and UHCMC)

# **VERSION NUMBER:**

Include the version number of this protocol if assigned by an outside entity.

DATE:

Click here to enter a date.

Objectives



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

# Directions: Describe the purpose, specific aims or objectives. Be sure to also include the hypothesis being tested

The AHA Stroke Rehabilitation guideline states that in the current fiscal climate, "the provision of comprehensive rehabilitation programs with adequate resources, dose, and duration is an essential aspect of stroke care and should be a priority" and recommends the development of "computeradapted assessments for personalized and tailored interventions" and "better predictor models to identify responders and non-responders" [1]. Patient baseline motor status and potential for motor recovery [2-12] should guide long-term rehabilitation goals. However, acute motor assessment and prognostication remain a clinically difficult task [13, 14]. Conventional clinical assessments (e.g. NIH Stroke Scale, Fugl-Meyer (FM) Scale) [15, 16] that power prognosis are highly dependent on the initial severity and care provider/point of care. In addition, those are often reduced further to even coarser prognostic scales (e.g. Orpington Prognostic Scale (OPS)) [17], which are limited due to ceiling effects, omission of fractionated and complex distal movements, and/or unequal weighting of the two extremities in assessments [18]. Furthermore, many survivors do not even receive comprehensive assessments prior to discharge. Besides, telestroke approaches implemented to address such issues are limited in their scope of care and still not fully developed for functional assessments [19-23]. This is critical because "all patients benefit from a formal assessment of the patient's rehabilitation needs prior to discharge" [24]. A simple portable technology that can holistically aid clinicians in: 1. detailed assessments of motor symptoms; 2. patient classification for rehabilitation; and 3. prediction of recovery, is lacking [12-14, 25-35].

We will investigate our Integrated sensor-based Motion Analysis Suite (IMAS) of motion capture cameras, force sensors, and inertial sensors, to objectively and quantitatively measure acute stroke patient motor status.

To this end, we will investigate one Specific Aim:

Aim 1: Assess the feasibility of using our IMAS for assessing acute stroke and predict outcome.

# Sub Aim 1.1: IMAS optimization and applicability in an acute stroke setting:

We hypothesize that it is possible to use an integrated set of sensors that can interface with acute or subacute stroke patients undergoing motor exams to extract features of their motor behavior. Thus, we will evaluate the feasibility of our IMAS prototype (with motion capture cameras, accelerometers, gyroscopes, and force sensors). For this purpose, we will assess the IMAS in acute or subacute ischemic or hemorrhagic stroke subjects subjects subjects subjects will undergo a series of IMAS upper limb focused tools such as FM, Barthel Index, and OPS assessments. We will also collect demographics, and stroke clinical information and imaging data from Magnetic Resonance (MRI)



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

# Background

Directions: Describe the relevant prior experience and gaps in current knowledge describing how it will add to existing knowledge. Include any relevant preliminary data.

The NIH National Institute of Neurological Disorders and Stroke (NINDS) sponsors this study It aims to investigate the feasibility of clinical use of an Integrated Motion Analysis Suite (IMAS) for stroke assessments. This technology is powered by software to objectively quantify stroke severity and predict stroke motor recovery.

Stroke is a leading cause of disability in the US, with ~6.5M survivors [37, 38]. Most survivors endure motor deficits (~70%) and require rehabilitation [1, 39-43]. Patient motor status and potential for recovery [2-12] should guide long-term rehabilitation goals. However, state-of-theart tools to predict the extent to which a patient can recover their motor abilities or even to measure current abilities are limited. In fact, many survivors do not even receive comprehensive assessments prior to discharge. Telestroke addresses such issues, yet is limited in its scope of care and still not fully developed for functional assessments [19-23]. This is critical because "all patients benefit from a formal assessment of the patient's rehabilitation needs prior to discharge" [24]. With an aging population, a projected 19% shortfall in US neurologists in the next 10 yrs. [44-47], and a lack of neurologists outside of metropolitan areas [48, 49] the problem is growing. Furthermore, conventional clinical assessments (e.g., NIH Stroke Scale, Fugl-Meyer (FM)) [15, 16] that power prognosis are highly dependent on the care provider/point of care and are often reduced to even coarser prognostic scales (e.g. Orpington Prognostic Scale (OPS)) [17]. These assessments help predict recovery potential and/or tailor rehabilitation. However, these tools are limited given ceiling effects, omission of fractionated and complex distal movements, and/or weighing the upper and lower limbs unequally [18, 50-52]. To address these limitations the AHA Stroke Rehabilitation guidelines specifically call for the development of "computer-adapted assessments for personalized and tailored interventions", "newer technologies such as... body-worn sensors", and "better predictor models to identify responders and non-responders" [1]. However, a simple technology that can holistically aid clinicians in: motor symptom assessments, patient classification, and prediction of recovery is lacking [12-14, 25-35].

Sensor-based measurements of movement kinematics/ kinetics quantify patient motor abilities (e.g., [53-64]). For example, wearable sensors and motion capture cameras offer highly portable options [53, 65-67] to assess motor performance and predict clinical scales [63, 68-70]. However, those are difficult to implement in clinical settings due to size, cost, and complexity [61, 71]). Another limitation pertains, their reliance on single sensor types/modalities or focus on specific joints and/or symptoms (and thus do not capture the systemic disease state) [53, 65-67].



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|



In summary, there is a great clinical need for a simple tool to assess stroke patient's motor abilities and predict likelihood of motor recovery. We will investigate a sensor-based system coupled with statistical algorithms to allow computational analysis of stroke injury, through data dimensionality reduction and prediction methods. This approach will provide the clinician with a tool to aid and augment the classic evaluation process.

# Inclusion and Exclusion Criteria

Describe how individuals will be screened for eligibility. Using the tables below, describe the inclusion and exclusion criteria that will define who will be included and excluded in your final study sample.

Recruited will take place at the following places:

- University Hospitals Cleveland Medical Center (UHCMC)
- 2. University of Illinois Hospital and Health System (UI Health)

Both of them have comprehensive neurology treatment and motor rehabilitation services available, including outstanding neurologists who can provide referrals of stroke patients to this study. We will invite those subjects deemed eligible to the lab for the consent process and an opportunity to ask additional questions. The research team will offer eligible patients enrollment in this study once confirmed safe and appropriate.

Information about patients who are not eligible will be shredded and not retained.

| | Inclusion Criteria |
|----|---------------------------------------------------------|
| 1. | Providing informed consent to participate in the study. |



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

| 2. | Age 18 to 85 years old. |
|---|---|
| 3. | Clinical presentation and neuroimaging (CTA-CTP/ MRI-MRA) consistent with the |
| | diagnosis of Acute Ischemic or Hemorrhagic Stroke [7, 93-97]. |
| 4. | Preserved mental status (Glasgow coma score >12: E(4), V(5), M (4-6)) [98] |
| 5. | Presence of upper limb weakness per the NIHSS (1-2 points in the arm) and ability to perform testing (i.e., NIHSS motor score 1-2 at elbow, wrist, and finger flexion-extension) [16, 99] within 30 days from stroke. (Note that individuals with a prior ischemic or hemorrhagic stroke with available information pertaining superior extremity baseline strength after their previous stroke would qualify). |
| 6. | Presence of upper limb weakness per the NIHSS (2 points in the arm) and ability to perform testing (i.e., NIHSS motor score 2 at elbow, wrist, and finger flexion-extension) [16, 99] in subacute stroke. (Note that individuals with a prior ischemic or hemorrhagic stroke with available information pertaining superior extremity baseline strength after their previous stroke would qualify). |
| 7. | Baseline Modified Rankin score <4 [100, 101]. |

| | Exclusion Criteria |
|---|---|
| 1. | History of dementia per relative/ medical records. |
| 2. | Presence of receptive aphasia at baseline or after the current acute stroke. |
| 3. | Need for rapid clinical response due to conditions such as psychosis, or suicidality. |
| 4. | Unstable medical conditions (e.g., uncontrolled diabetes, uncompensated cardiac issues, heart failure, pulmonary issues, or chronic obstructive pulmonary disease);" |
| 5. | Amputated limbs [16, 99]. |
| 6. | Absence of weakness as per the NIHSS (0 points = no drift for motor arm and leg items) or severe motor impairment NIHSS 4 points for motor arm)[16, 99]. |
| 7. | Stroke mimics (e.g., infections, medication effects from sedatives, electrolyte imbalances, etc.). |
| 8. | Stroke worsening between assessments. |

# Number of Research Participants

Directions: Indicate the target number of research participants to be accrued locally, and, if this is a multi-site study, indicate the total number of research participants to be accrued across all sites.

Up to 60 patients with a diagnosis of stroke, and meeting the above criteria will be recruited on both following sites.

- 1. University Hospitals Cleveland Medical Center
- 2. University of Illinois Hospital and Health System
- 3. Sinai Chicago Medical Center (affiliated to Schwabb Rehabilitation Medical Center)

# Recruitment Methods



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

Describe how subjects will be identified (the source of potential research participants), and also how, when, and where they will be recruited. Describe all methods of contact / communication.

We will recruit up to 60 subjects for this study, with the intention of enrolling exactly 30 subjects with stroke to account for screen failures and withdrawals of subjects (e.g., some of the patients who are recruited and pre-screened into the study might worsen or fluctuate and then would be excluded following previous visits).

Potential subjects will be identified by the following sources:

- 1. Attending physicians or therapists may refer their patients to the study.
- 2. Via the UHCMC and UI Health inpatient facilities.
- 3. Possible subjects might also be identified through their medical records and their physicians might be asked to inform the subject about the study.

We anticipate that subjects will be primarily recruited through the University Hospitals Cleveland Medical Center and University of Illinois Hospital and Health System. All patients receiving inpatient care for stroke at University Hospitals Cleveland Medical Center and University of Illinois Hospital and Health System will be eligible for this study. We will also approach colleagues at the other collaborating teaching hospitals and institutions in the greater Cleveland area and Chicago area. Overall, we anticipate a large population with stroke that will be eligible for this study allowing for the effective recruitment of 30 patients.

Eligible patients will be offered enrollment in this study once deemed safe and appropriate by the research team.

Informed consent will be obtained by the study PI and/or a co-investigator in person. The test procedures will be described and the testing equipment will be shown to the subject. Study co-investigators will clearly explain all the procedures and risks of the testing outlined in the consent form. The subject will be given the time needed to consider their decision and will be encouraged to ask questions, both during the initial interview and throughout the study. The PI or a co-investigator will answer any questions regarding the study at the time consent is given. Once enrolled, the subject may pause or terminate his/her participation at any time during the study.

Retention of subjects is feasible, particularly because of the facilities available at the University Hospitals Cleveland Medical Center, which is a top hospital with Comprehensive Stroke Center Certification (Honor Roll Elite Plus Gold Plus status) and University of Illinois Hospital and Health System designed to promote accessibility for a diverse population of patients with mobility issues. Patient retention will be encouraged/ followed by study staff via communication with the patients throughout the research study, such as to check in on patients and help arrange transportation to the medical center.

Patients will also be compensated for their time and effort as detailed in the section below.

#### Setting

All research related activities in this protocol will be performed at the main University Hospitals Cleveland Medical Center and University of Illinois Hospital and Health System facility. Recruitment



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

of potential participants would be carried out from the inpatient facilities (preferentially Lerner Tower 4th floor) at University Hospitals Cleveland Medical Center at 11100 Euclid Avenue. For University Hospitals Cleveland Medical Center facility, research procedures will occur inside the laboratory of the DCRU. For University of Illinois Hospital and Health System, research procedures will occur at the following locations:

- 1. 1740 W Taylor Street, Suite C-100 M/C889, Chicago IL 60612
- 2. 1801 W Taylor Street, room 1307, 1320 or 1314A, Chicago IL 60612

#### Consent Process

This study will be obtaining consent but request a partial waiver of HIPAA authorization for screening purposes. Specifically, we would like to collect limited information from the medical record directly pertaining eligibility information about potential subjects from the medical record (i.e., diagnosis of stroke and other information pertaining to inclusion/exclusion criteria). Individuals with a prior ischemic or hemorrhagic stroke with available information pertaining superior extremity baseline strength after their previous stroke. The research team may contact the patients' caregivers to gather this information to ascertain their eligibility to enter the study.

Sharing of Results with Research Participants

- Results will <u>not</u> be shared with research participants
- ☐ Results will <u>not</u> be shared with research participants' doctors

#### Study Design

This study will have 1 screening visit and 5 evaluation visits and use a battery of sensors for acquiring patent movement kinematic and kinetic data.

We will recruit up to 60 subjects for this study, with the intention of enrolling exactly 30 subjects with stroke to account for screen failures and withdrawals of subjects (e.g., some of the patients who are recruited and pre-screened into the study might worsen or fluctuate and then would be excluded following previous visits).

#### Study Procedures

#### <u>Pre-screening Procedures:</u>

During the pre-screening process, the investigators will approach the clinical stroke care team to learn about potential candidates admitted with acute or subacute stroke in the privacy of the Stroke team's work room ("Fishbowl") at Lerner Tower 4<sup>th</sup> Floor at UHCMC or other approved facilities. For University of Illinois Hospital and Health System, research procedures will occur at the following locations:

- 1. 1740 W Taylor Street, Suite C-100 M/C889, Chicago IL 60612
- 2. 1801 W Taylor Street, room 1307, 1320 or 1314A, Chicago IL 60612

Once this information is collected, the coordinator will consult with the principal investigator, who will then give approval for the subject to be screened. The pre-screening process will last duration of approximately 15'.



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

# Screening

(Approximate Time: 20 mins)

# Screening Procedures:

At Screening the PI and the co-investigators will conduct a review of inclusion/exclusion criteria to determine the subject's eligibility for enrollment. Study procedures will be reviewed with the subject, and documentation of informed consent will be obtained.

At Screening the following procedures will be completed:

- Discuss study-specific procedures with the subject.
- Review inclusion and exclusion criteria.
- PI will review the initial assessment of the subjects to determine which subjects have a diagnosis of stroke.
- Obtain a signed and dated consent form.
- Patient demographics and medical information obtained from Medical records such as collection of stroke lesion information from MRI, collection of time from stroke onset information, etc.

# Evaluation 1

Initial Evaluation - (Approximate Time: 90')

This visit might be completed on the same day as the screening visit if time allows and it is convenient for the subject.

- Fugl-Meyer evaluation
- OPS evaluation
- Barthel Index evaluation



Adverse events NIH-CDE questionnaire

Note, all patients will undergo stroke standardized multidisciplinary rehabilitation (independent of these experiments).

# Evaluations 2-4

Evaluation - (Approximate Time: 90')

These visits will be scheduled in acute or subacute strokes in the wards and other approved testing areas.

During each visit, the subject will complete a series of assessments:

Adverse events NIH-CDE questionnaire.

#### Evaluation 5



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

This visit will be scheduled after rehabilitation completion (during a standard clinic follow-up). All patients will receive standard physical and/or occupational therapy as indicated by our PT specialists and followed by standardized exercises for home therapy as needed.

Final Evaluation (5) - (Approximate Time: 90 mins)

- Fugl-Meyer evaluation
- OPS evaluation
- Barthel Index evaluation
- Adverse events NIH-CDE questionnaire.

We will perform up to 4 assessments in the initial phase and then 1 follow up. Subjects will be asked before each 90-minute research session whether they feel up to completing the physical study activities, and also that the study team will verify before the session with nursing that the research session does not conflict with any clinical care, e.g., MRI or therapy session.

#### DESCRIPTION OF ASSESSMENTS:

A research team member will conduct the following assessments:

Fugl-Meyer (FM): We will conduct a FM assessment (upper limb) [15]. The FM score is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment. There are no associated risks with these measures and do not add any more stress than standard physical movements. If subject's become fatigued they will be informed they can take a break at any point during the assessment.

Orpington Prognostic Scale (OPS): We will conduct an OPS assessment [102]. The OPS is an assessment of stroke severity (e.g., motor deficits, proprioception, balance and cognition). It is applied clinically and in research. There are no associated risks with these measures and do not add any more stress than standard physical movements. If subject's become fatigued they will be informed they can take a break at any point during the assessment.

Barthel Index: We will conduct a Barthel Index assessment[100]. The Barthel Index questionnaire measures the extent to which somebody can function independently and has mobility in their activities of daily living (ADL) i.e., feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. The index also indicates the need for assistance in care. The BI is a widely used measure of functional disability. There are no associated risks with these measures.



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|



These assessments do not add any more stress than standard physical movements. If subjects become fatigued, they will be informed they can take a break at any point during the assessment. During motion tasks patients will not be asked to perform movements that they feel they are incapable of performing or cause excessive stress. Assessments will be made during the neurological examination of the patient (partly to gather data to determine the FM information), and no added risks will be made beyond what is seen in a typical neuro/motor exam. During motion tasks patients will not be asked to perform movements that they feel they are incapable of performing or cause excessive stress. Assessments include:



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|



Data to be Collected for your study (AFTER consent and HIPAA Authorization have been obtained)

List all data to be collected for the research study or attach a data collection sheet (e.g. laboratory values, physician notes, length of stay, etc.)

Also, the following data will be collected:

- Telephone number
- Email address
- Address
- Medical record number



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

- Dates related to an individual (e.g., date of admission, birth, surgery, etc)
- Name
- PMH
- Imaging Data
- OPS
- Barthel Index

# Data Analysis Plan

after rehabilitation.

We determined the sample size (recruitment up to 60 subjects for n=30 subjects completing the protocol) based on: 1. A sample size of N=15 patients provides at least 80% power (alpha=0.05) to detect a mean difference of 3% in arm movement mean speed, 2.7% in arm movement mean peak speed, and 2.5% in arm movement jerk between an affected and non-affected limb.





| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

Data forms and questionnaires: we will code those in a standardized manner, and enter them into our database. We will track and regularly back up digital measures/recordings in our database. Analyses will involve the use of standard statistical software such as R and MATLAB.

# Confidentiality

To ensure confidentiality we will:

- Use a unique study identifier (not derived from the participants personal identifiers) to code individuals' data and I will store this ID log separate from study data.
- Store the electronic data in a UH Secure Network Drive for UHCMC and UIC Secure Network Drive for UI Health.
- Store paper research data and documents in locked secure environment safe-locked cabinet.
   For UHCMC, room#108, 2027 Cornell Road, Cleveland, OH 44106. For UI Health 1801 W.
   Taylor St., room 1309, Chicago IL 60612.
- De-identified patient data will be shared with the other collaborators on this NIH study. This
  data involves results from our testing.

#### As for HIPAA Authorization:

- We are requesting a full or partial waiver of HIPAA for prescreening
- Note, this study requires access to protected health information about patients prior to their
  consent to assess eligibility for potential participation. Their PHI might come from electronic
  or paper file medical record access or by way of the healthcare providers' personal knowledge
  of the patients' health information. Specifically, to collect eligibility information about
  potential subjects from the medical record such as whether a person or persons have stroke,
  and other inclusion and exclusion criteria.
- We will keep any potential identifiers for 3 years beyond the conclusion of present study's procedures, data collection and analysis.
- PHI collected for purposes of this research study will not be reused or disclosed to any other
  person or entity, except as required by law, for authorized oversight of the research study, or
  for other research for which the use of disclosure of protected health information for which
  an authorization or opportunity to agree or object is not required by 45 CFR 164.512.

#### Risks to Research Participants

List the reasonably foreseeable risks such as breach of confidentiality, discomforts, hazards, or inconveniences to the research participants related to their participation in the research. Include a description of the probability, magnitude, duration, and reversibility of the risks. Include the physical psychological, social, legal, and economic risks.

#### Questionnaires and motor assessments:

There are potential risks of personal discomfort to answer the questionnaires.

There are some potential risks of fall, syncope and fatigue posed to subjects during recording of data with the biomechanical sensor suite. We will make sure that our study team will stand near the subjects



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

so that we can provide support at any time. If participants become fatigued during testing or are uncomfortable answering any personal questions, they will be informed that they are allowed to take a break at any point during the experiment and that they may end their participation at any time.

# Risk of breach of confidentiality

There is a risk of breach of confidentiality because someone who is not a part of the research team involved with this study might view your data either by accident or from malicious actions they take to hack the data. We are protecting against this possibility by only storing information that can be directly linked to you on UH computers, in password-protected files, which are behind firewalls.

# Provisions to Protect the Privacy Interests of Research Participants

Directions: Describe the steps that will be taken to protect research participants' privacy interests. (Consider issues such as physical space, proximity to other, and participant preferences)

For University Hospitals Cleveland Medical Center facility, screening, consenting and any research interventions will occur in private patient care rooms at the UHCMC inpatient facilities (Lerner Tower 4<sup>th</sup> floor). For UI Health, screening, consenting and any research interventions will occur in private patient care rooms at the following locations:

- 1. 1740 W Taylor Street, Suite C-100 M/C889, Chicago IL 60612
- 2. 1801 W Taylor Street, room 1307, 1320 or 1314A, Chicago IL 60612

#### Potential Benefit to Research Participants

Describe the potential benefits that individual research participants may experience from taking part in the research. Include the probability, magnitude, and duration of the potential benefits. If there is no direct benefit, state the potential benefit to society.

There is no direct benefit to subjects for participating in this research study.

However, stroke is a serious issue, particularly in an older adult population. Thus, a benefit for society overall is related to addressing the pressing need for stroke prognosis.

# Withdrawal of Research Participants

Directions: Describe the anticipated circumstances under which research participants will be withdrawn from the research without their consent. Also include the procedures that will be followed when a research participant withdraws or are withdrawn from the research, including partial withdrawal from procedures with continued data collection.

The study doctor will inform the participants about new information or changes in the study that may affect their health or willingness to continue in the study. The study staff may take the participant out of the study without its permission if any of the following occurred:

- If there are subject health changes and the study is no longer in subject best interest



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

- If new information becomes available that warrants stopping participation
- If the participant does not follow the study requirements
- If the study is stopped by the sponsor, Institutional Review Board (IRB).

If any of these events occurred, the study doctor will explain why the subject needs to stop taking part in the study. We will also talk to the participant about follow-up care if needed. If the subject withdraws from the study prior to its completion for any reason, we will request a final clinical visit to ensure subject safety. In the event that further care is needed, the research team will direct the subject to the appropriate resources. If a subject decided to stop participating, it may decide whether or not to let the study doctor continue to provide its medical information to the organization running the study.

# Alternatives to Participation

Directions: List other available clinical treatments, what would be included if a subject continued on standard of care therapy. If this is not a clinical trial, you may select the box indicating that the alternative is not to participate. If there is a viable alternative you must list it in the consent.

This is not a clinical trial. Subjects alternative is not to participate.

# Costs to Research Participants

Describe what costs research participants will be responsible for as a result of their participation in the research, including but not limited to: clinical services required by the protocol deemed billable to insurance, transportation to study visits, parking, costs of drugs, cost of therapy, lost broken or stolen devices, etc. Explain who will be responsible for payment of provided services in the event of insurance denials. List what procedures, drugs, devices, supplies will be paid by the study sponsor or covered by other funding. List the other funding source.

There are no costs to research participants or their insurance companies.

# Research Participant Compensation

Describe the schedule, payment method, and payment total of any incentives or compensation that research participants will receive for participation in the research (e.g., gift cards or cash with amount, t-shirts, devices, bags, swag, etc.)

Describe the schedule, payment method, and payment total of any reimbursement that research participants will receive for participation in the research (e.g., gift cards or cash with amount, etc.)

Subjects will receive \$25/visit or evaluation, which means subjects will be compensated \$50 for the day that has 2 evaluations. Study funds will also cover the cost of parking (in the Rainbow parking garage) for evaluation 5. Additional transportation costs will be reviewed by the study PI and may be redeemed on a case-by-case basis.

Funding agency is not providing any payment for injury.

Provisions to Monitor the Data to Ensure the Safety of Research Participants

Describe how often the data will be monitored for completeness, accuracy and adherence to the protocol.



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

Indicate if there will be a Data and Safety Monitoring Board or Committee. Provide information about the DSMB/C including the contact information of the committee member(s) (as applicable); whether it is independent from the study sponsor; how often it meets; the type of data that will be used; written reports, etc.

We will review adverse events following each patient visit. All adverse events, regardless of attribution to evaluation with the motor analysis suite, will be collected and recorded, using standard adverse event forms. A diagnosis, rather than signs, symptoms, and/or other clinical information, will be recorded when possible. Subjects will be asked in an open-ended manner about the presence of any adverse events. We will assess adverse events per the NIH CDE instrument. All applicable local regulatory requirements related to serious adverse events will be followed during this study. Serious adverse events will be promptly reported to the IRB, the General Clinical Research Center, the NIH. The issue of placing the study on hold will be raised by the investigators with our local IRB if any serious adverse events occur.

The PI or study staff will review all data collection forms on an ongoing basis for data completeness and accuracy as well as protocol compliance. Data collected will be reviewed by a member of study staff not responsible for the collection of that data set.

# Drugs or Devices

No drugs or devices will be used interventionally for this research project.

#### Additional Information

Directions: If you have any additional information regarding your study not covered in the template, please include it here.

Upon receiving funding, a research fellow and research nurse support through the Dahm's unit will be added to the protocol per the NIH budget that was submitted.

#### Community-Based Participatory Research

Describe the involvement of the community in the design and conduct of the research.

Note: Community based research is research that is conducted as an equal partnership between academic investigators and members of a community. In Community Based Participatory Research (CBPR) protects, the community participates fully in all aspects of the research process.

This is not a community-based participatory research project.

#### International information

If you will be conducting international research, address the following issues:

- Sites/locations
- Data sharing

This is not an international study.

#### References



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

Please reference the Investigator Manual for local institutional requirements.

- Winstein, C.J., et al., Guidelines for Adult Stroke Rehabilitation and Recovery. A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association, 2016.
- 2. Hommel, M., et al., Social dysfunctioning after mild to moderate first-ever stroke at vocational age. J Neurol Neurosurg Psychiatry, 2009. 80(4): p. 371-5.
- 3. Brown, D.L., et al., Projected costs of ischemic stroke in the United States. Neurology, 2006. 67(8): p. 1390-5.
- 4. Lindenberg, R., et al., Structural integrity of corticospinal motor fibers predicts motor impairment in chronic stroke. Neurology, 2010. 74(4): p. 280-7.
- 5. Werring, D., et al., Diffusion tensor imaging can detect and quantify corticospinal. J Neurol Neurosurg Psychiatry, 2000. 69(2): p. 269-72.
- 6. Maraka, S., et al., Degree of corticospinal tract damage correlates with motor function after stroke. Ann Clin Transl Neurol, 2014. 1(11): p. 891-9.
- 7. Fritz, S.L., et al., Active finger extension predicts outcomes after constraint-induced movement therapy for individuals with hemiparesis after stroke. Stroke, 2005. 36(6): p. 1172-
- 8. Wolf, S.L., et al., The EXCITE trial: attributes of the Wolf Motor Function Test in patients with subacute stroke. Neurorehabil Neural Repair, 2005. 19(3): p. 194-205.
- 9. Fries, W., A. Danek, and T.N. Witt, Motor responses after transcranial electrical stimulation of cerebral hemispheres with a degenerated pyramidal tract. Ann Neurol, 1991. 29(6): p. 646-50.
- 10. Lang, C.E. and M.H. Schieber, Human finger independence: limitations due to passive mechanical coupling versus active neuromuscular control. J Neurophysiol, 2004. 92(5): p. 2802-10.
- 11. Kuypers, H.G.J.M., A New Look at the Organization of the Motor System. Progress in Brain Research, 1982. 57: p. 381-403.
- 12. Veerbeek, J.M., et al., Early Prediction of Outcome of Activities of Daily Living After Stroke. A Systematic Review, 2011. 42(5): p. 1482-1488.
- 13. Heinemann, A.W., et al., Prediction of rehabilitation outcomes with disability measures. Arch Phys Med Rehabil, 1994. 75(2): p. 133-43.
- 14. Saposnik, G., The Art of Estimating Outcomes and Treating Patients With Stroke in the 21st Century. Stroke, 2014. 45(6): p. 1603-1605.
- 15. Fugl-Meyer, A.R., et al., The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med, 1975. 7(1): p. 13-31.
- Spilker, J., et al., Using the NIH Stroke Scale to assess stroke patients. The NINDS rt-PA Stroke Study Group. J Neurosci Nurs, 1997. 29(6): p. 384-92.
- 17. Rieck, M. and J. Moreland, The Orpington Prognostic Scale for patients with stroke: reliability and pilot predictive data for discharge destination and therapeutic services. Disabil Rehabil, 2005. 27(23): p. 1425-33.



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

- 18. Gladstone, D.J., C.J. Danells, and S.E. Black, The fugl-meyer assessment of motor recovery after stroke: a critical review of its measurement properties. Neurorehabil Neural Repair, 2002. 16(3): p. 232-40.
- 19. Akbik, F. and T.M. Leslie-Mazwi, The State of Telestroke. Endovascular Today, 2017. Feb 2017.
- Wechsler, L.R., et al., Telemedicine Quality and Outcomes in Stroke: A Scientific Statement for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke, 2017. 48(1): p. e3-e25.
- 21. Silva, G.S., et al., The status of telestroke in the United States: a survey of currently active stroke telemedicine programs. Stroke, 2012. 43(8): p. 2078-85.
- 22. Leira, E.C., et al., The growing shortage of vascular neurologists in the era of health reform: planning is brain! Stroke, 2013. 44(3): p. 822-7.
- 23. Commission, T.J., National Patieint Safety Goals. 2018.
- 24. Prvu Bettger, J.A., et al., Assessing stroke patients for rehabilitation during the acute hospitalization: findings from the get with the guidelines-stroke program. Arch Phys Med Rehabil, 2013. 94(1): p. 38-45.
- 25. Korner-Bitensky, N., et al., Motor and functional recovery after stroke: accuracy of physical therapists' predictions. Arch Phys Med Rehabil, 1989. 70(2): p. 95-9.
- 26. Allen, C., Predicting the outcome of acute stroke: a prognostic score. Journal of Neurology, Neurosurgery & Psychiatry, 1984. 47(5): p. 475-480.
- 27. Burke Quinlan, E., et al., Neural function, injury, and stroke subtype predict treatment gains after stroke. Ann Neurol, 2015. 77(1): p. 132-45.
- Lai, S.M., P.W. Duncan, and J. Keighley, Prediction of functional outcome after stroke: comparison of the Orpington Prognostic Scale and the NIH Stroke Scale. Stroke, 1998. 29(9): p. 1838-42.
- Hendricks, H., et al., Motor Recovery after Stroke: A systematic Review of the Literature.
   Vol. 83. 2002. 1629-37.
- 30. Langhorne, P., F. Coupar, and A. Pollock, Motor recovery after stroke: a systematic review. Lancet Neurol, 2009. 8(8): p. 741-54.
- 31. Chen, Z., et al., Evaluating ischemic stroke with diffusion tensor imaging. Neurol Res, 2008. 30(7): p. 720-6.
- 32. Weimar, C., et al., Predicting functional outcome and survival after acute ischemic stroke. J Neurol, 2002. 249(7): p. 888-95.
- 33. Macciocchi, S.N., et al., Ischemic stroke: relation of age, lesion location, and initial neurologic deficit to functional outcome. Arch Phys Med Rehabil, 1998. 79(10): p. 1255-7.
- 34. Kelly, P.J., et al., Functional recovery following rehabilitation after hemorrhagic and ischemic stroke. Arch Phys Med Rehabil, 2003. 84(7): p. 968-72.
- 35. Stinear, C.M., et al., The PREP algorithm predicts potential for upper limb recovery after stroke. Brain, 2012. 135(Pt 8): p. 2527-35.
- 36. Coleman, E.R., et al., Early Rehabilitation After Stroke: a Narrative Review. Curr Atheroscler Rep, 2017. 19(12): p. 59.
- 37. Mozaffarian, D., et al., Heart Disease and Stroke Statistics—2016 Update. A Report From the American Heart Association, 2015.



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

- 38. Bronnum-Hansen, H., et al., Long-term survival and causes of death after stroke. Stroke, 2001. 32(9): p. 2131-6.
- 39. Kwakkel, G., et al., Probability of regaining dexterity in the flaccid upper limb: impact of severity of paresis and time since onset in acute stroke. Stroke, 2003. 34(9): p. 2181-6.
- 40. Hankey, G.J., et al., Long-term disability after first-ever stroke and related prognostic factors in the Perth Community Stroke Study, 1989-1990. Stroke, 2002. 33(4): p. 1034-40.
- 41. Takeuchi, N. and S. Izumi, Rehabilitation with poststroke motor recovery: a review with a focus on neural plasticity. Stroke Res Treat, 2013. 2013: p. 128641.
- 42. Gadidi, V., et al., Long-term outcome poststroke: predictors of activity limitation and participation restriction. Archives of physical medicine and rehabilitation, 2011. 92(11): p. 1802-1808.
- 43. Writing Group, M., et al., Heart disease and stroke statistics--2010 update: a report from the American Heart Association. Circulation, 2010. 121(7): p. e46-e215.
- 44. Dall, T.M., et al., Supply and demand analysis of the current and future US neurology workforce. Neurology, 2013. 81(5): p. 470-8.
- 45. IHS and A.o.A.M. Colleges, The Complexities of Physician Supply and Demand: Projections from 2013 to 2025 (prepared for the Association of American Medical Colleges). 2015. p. 68.
- 46. Harrah, S., Beyond Primary Care: Which Specialties Are Needed in Growing Physician Shortage. University of Medicine and Health Sciences (UMHS) News, 2014. Obamacare, Primary Care, Residency News, U.S. Doctor Shortage.
- 47. Freeman, W.D., et al., The Workforce Task Force report: clinical implications for neurology. Neurology, 2013. 81(5): p. 479-86.
- 48. (AAN), A.A.o.N., Neurology Workforce Data.
- 49. Shih, L.C., D. Tarsy, and M.S. Okun, The current state and needs of north american movement disorders fellowship programs. Parkinsons Dis, 2013. 2013: p. 701426.
- 50. Pandian, S. and K.N. Arya, Stroke-related motor outcome measures: do they quantify the neurophysiological aspects of upper extremity recovery? J Bodyw Mov Ther, 2014. 18(3): p. 412-23.
- 51. Harrison, J.K., K.S. McArthur, and T.J. Quinn, Assessment scales in stroke: clinimetric and clinical considerations. Clin Interv Aging, 2013. 8: p. 201-11.
- 52. Orgogozo, J.M., Advantages and disadvantages of neurological scales. Cerebrovasc Dis, 1998. 8 Suppl 2: p. 2-7.
- 53. Patel, S., et al., A review of wearable sensors and systems with application in rehabilitation. J Neuroeng Rehabil, 2012. 9: p. 21.
- 54. Alt Murphy, M.H., C.K., Kinematic analysis of the upper extremity after stroke how far have we reached and what have we grasped? Physical Therapy Reviews 2015. 20(3): p. 137-155.
- 55. DeJong, S.L., S.Y. Schaefer, and C.E. Lang, Need for speed: better movement quality during faster task performance after stroke. Neurorehabil Neural Repair, 2012. 26(4): p. 362-73.
- 56. Alt Murphy, M., C. Willen, and K.S. Sunnerhagen, Kinematic variables quantifying upper-extremity performance after stroke during reaching and drinking from a glass. Neurorehabil Neural Repair, 2011. 25(1): p. 71-80.



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

- 57. Aprile, I., et al., Kinematic analysis of the upper limb motor strategies in stroke patients as a tool towards advanced neurorehabilitation strategies: a preliminary study. Biomed Res Int, 2014. 2014: p. 636123.
- 58. Silva, R.M.S., E.; Fonseca, P.; Pinheiro, A.R.; Silva, C.; Correia, M.V.; Mouta, S., Analysis and Quantification of Upper-Limb Movement in Motor Rehabilitation After Stroke, in Biosystems & Biorobotics book series (BIOSYSROB\_. 2016.
- 59. Cirstea, M.C. and M.F. Levin, Compensatory strategies for reaching in stroke. Brain, 2000. 123 (Pt 5): p. 940-53.
- 60. Bigoni, M., et al., Does kinematics add meaningful information to clinical assessment in post-stroke upper limb rehabilitation? A case report. J Phys Ther Sci, 2016. 28(8): p. 2408-13.
- 61. Reinkensmeyer, D.J., et al., Computational neurorehabilitation: modeling plasticity and learning to predict recovery. J Neuroeng Rehabil, 2016. 13(1): p. 42.
- 62. Dipietro, L., et al., Learning, not adaptation, characterizes stroke motor recovery: evidence from kinematic changes induced by robot-assisted therapy in trained and untrained task in the same workspace. IEEE Trans Neural Syst Rehabil Eng, 2012. 20(1): p. 48-57.
- 63. Volpe, B.T., et al., Robotic devices as therapeutic and diagnostic tools for stroke recovery. Arch Neurol, 2009. 66(9): p. 1086-90.
- 64. Dipietro, L., et al., Submovement changes characterize generalization of motor recovery after stroke. Cortex, 2009. 45(3): p. 318-24.
- 65. Bonato, P., Clinical applications of wearable technology. Conf Proc IEEE Eng Med Biol Soc, 2009. 2009: p. 6580-3.
- 66. Del Din, S., et al., Estimating Fugl-Meyer clinical scores in stroke survivors using wearable sensors. Conf Proc IEEE Eng Med Biol Soc, 2011. 2011: p. 5839-42.
- 67. Patel, S., et al., Tracking motor recovery in stroke survivors undergoing rehabilitation using wearable technology. Conf Proc IEEE Eng Med Biol Soc, 2010. 2010: p. 6858-61.
- 68. Tran, V.D., P. Dario, and S. Mazzoleni, Kinematic measures for upper limb robot-assisted therapy following stroke and correlations with clinical outcome measures: A review. Med Eng Phys, 2018. 53: p. 13-31.
- 69. Krebs, H.I., et al., Robotic measurement of arm movements after stroke establishes biomarkers of motor recovery. Stroke, 2014. 45(1): p. 200-4.
- 70. Bosecker, C., et al., Kinematic robot-based evaluation scales and clinical counterparts to measure upper limb motor performance in patients with chronic stroke. Neurorehabil Neural Repair, 2010. 24(1): p. 62-9.
- 71. Chen, C.C. and R.K. Bode, Factors influencing therapists' decision-making in the acceptance of new technology devices in stroke rehabilitation. Am J Phys Med Rehabil, 2011. 90(5): p. 415-25.
- 72. Robertson, D.G.E., et al., Research Methods in Biomechanics. 2013.
- 73. Jenkins, S.P.R., Sports Science Handbook. Vol. 1: A-H. 2005, Great Britain: Multi-Science Publishing Co. Ltd.
- 74. Mancini, M., et al., ISway: a sensitive, valid and reliable measure of postural control. J Neuroeng Rehabil, 2012. 9: p. 59.
- 75. Headon, R. and R. Curwen. Recognizing movements from the ground reaction force. in PUI '01 Proceedings of the 2001 workshop on Perceptive user interfaces 2001.



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

- 76. Richards, J.G., The measurement of human motion: A comparison of commercially available systems. Human Movement Science, 1999. 18: p. 589-602.
- 77. Bartlett, R., Introduction to Sport Biomechanics. 2007, New York: Routledge, Taylor & Francis Group.
- 78. Chen, X. and J. Davis, Camera Placement Considering Occlusion for Robust Motion Capture, in Stanford Computer Science Technical Report. 2000, Stanford.
- 79. Szczerbik, E. and M. Kalinowska, The influence of knee marker placement error on evaluation of gait kinematic parameters. Acta Bioeng Biomech, 2011. 13(3): p. 43-6.
- 80. Ran, Y., et al., Applications of a simple characterization of human gait in surveillance. IEEE Trans Syst Man Cybern B Cybern, 2010. 40(4): p. 1009-20.
- 81. Sturm, P.F., Critical Motion Sequences for the Self-Calibration of Cameras and Stereo Systems with Variable Focal Length. Image and Vision Computing, 2002. 20(5-6): p. 415-426.
- 82. Pourcelot, P., et al., A method to synchronise cameras using the direct linear transformation technique. J Biomech, 2000. 33(12): p. 1751-4.
- 83. N.R. Miller, R. Shapiro, and T.M. McLaughlin, A technique for obtaining spatial kinematic parameters of segments of biomechanical systems from cinematographic data. J Biomechanics, 1980. 13(535-547).
- 84. Milner, C.E., Motion analysis using online systems, in Biomechanical Analysis of Movement in Sport and Exercise: the British Association of Movement in Sport and Exercise Sciences Guide. 2007, Oxon: Routledge.
- 85. Perez-Sala, X., et al., A survey on model based approaches for 2D and 3D visual human pose recovery. Sensors (Basel), 2014. 14(3): p. 4189-210.
- 86. Papapetropoulos, S., et al., Objective quantification of neuromotor symptoms in Parkinson's disease: implementation of a portable, computerized measurement tool. Parkinsons Dis, 2010. 2010: p. 760196.
- 87. Lun, R. and W. Zhao, A Survey of Applications and Human Motion Recognition with Microsoft Kinect. International Journal of Pattern Recognition and Artificial Intelligence, 2015. 29(5).
- 88. Berger, K., et al., A State of the Art Report on Kinect Sensor Setups in Computer Vision, in Lecture Notes in Computer Science., M. Grzegorzek, et al., Editors. 2013, Springer Berlin Heidelberg. p. 257–272.
- 89. Schepers, M., Ambulatory Assessment of Human Body Kinematics and Kinetics. 2009, Universiteit Twente: Netherlands. p. 148.
- 90. Rocchi, L., L. Chiari, and F.B. Horak, Effects of deep brain stimulation and levodopa on postural sway in Parkinson's disease. J Neurol Neurosurg Psychiatry, 2002. 73(3): p. 267-74.
- 91. Taylor-Rowan, M., et al., Functional Assessment for Acute Stroke Trials: Properties, Analysis, and Application. Front Neurol, 2018. 9: p. 191.
- 92. Stinear, C.M., et al., Functional potential in chronic stroke patients depends on corticospinal tract integrity. Brain, 2007. 130(Pt 1): p. 170-80.
- 93. Jauch, E.C., et al., Guidelines for the early management of patients with acute ischemic stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke, 2013. 44(3): p. 870-947.



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

- 94. Allen, L.M., et al., Sequence-specific MR imaging findings that are useful in dating ischemic stroke. Radiographics, 2012. 32(5): p. 1285-97; discussion 1297-9.
- 95. Siddiqui, F.M., S.V. Bekker, and A.I. Qureshi, Neuroimaging of hemorrhage and vascular defects. Neurotherapeutics, 2011. 8(1): p. 28-38.
- 96. Kang, B.K., et al., Diffusion-weighted MR imaging of intracerebral hemorrhage. Korean J Radiol, 2001. 2(4): p. 183-91.
- 97. Smania, N., et al., Active finger extension: a simple movement predicting recovery of arm function in patients with acute stroke. Stroke, 2007. 38(3): p. 1088-90.
- 98. Teasdale, G. and B. Jennett, Assessment of coma and impaired consciousness. A practical scale. Lancet, 1974. 2(7872): p. 81-4.
- 99. NIH. NIH Stroke Scale. Available from: <a href="http://www.strokecenter.org/wp-content/uploads/2011/08/NIH">http://www.strokecenter.org/wp-content/uploads/2011/08/NIH</a> Stroke Scale.pdf.
- 100. Sulter, G., C. Steen, and J. De Keyser, Use of the Barthel index and modified Rankin scale in acute stroke trials. Stroke, 1999. 30(8): p. 1538-41.
- Banks, J.L. and C.A. Marotta, Outcomes validity and reliability of the modified Rankin scale: implications for stroke clinical trials: a literature review and synthesis. Stroke, 2007. 38(3): p. 1091-6.
- 102. Pittock, S.J., et al., The Orpington Prognostic Scale within the first 48 hours of admission as a predictor of outcome in ischemic stroke. J Stroke Cerebrovasc Dis, 2003. 12(4): p. 175-81.
- 103. Han, J., et al., Enhanced computer vision with microsoft kinect sensor: A review. IEEE Trans. Cybern., 2013 43(5): p. 1318–1334.
- 104. Khasnis, A. and R.M. Gokula, Romberg's test. J Postgrad Med, 2003. 49(2): p. 169-72.
- 105. Jankovic, J., Parkinson's disease: clinical features and diagnosis. J Neurol Neurosurg Psychiatry, 2008. 79(4): p. 368-76.
- 106. Arciniegas, D.B., C.A. Anderson, and C.M. Filley, Behavioral Neurology & Neuropsychiatry. 2013, New York: Cambridge University Press.
- 107. Goetz, C.G., et al., Teaching tape for the motor section of the unified Parkinson's disease rating scale. Mov Disord, 1995. 10(3): p. 263-6.
- 108. Stinear, C.M., et al., Predicting Recovery Potential for Individual Stroke Patients Increases Rehabilitation Efficiency. Stroke, 2017. 48(4): p. 1011-1019.
- 109. Stinear, C.M., W.D. Byblow, and S.H. Ward, An update on predicting motor recovery after stroke. Ann Phys Rehabil Med, 2014. 57(8): p. 489-98.
- 110. Dipietro, L., et al., Changing motor synergies in chronic stroke. J Neurophysiol, 2007. 98(2): p. 757-68.
- 111. Dipietro, L., A.M. Sabatini, and P. Dario, Artificial neural network model of the mapping between electromyographic activation and trajectory patterns in free-arm movements. Med Biol Eng Comput, 2003. 41(2): p. 124-32.
- 112. Finley, M.A., et al., The effect of repeated measurements using an upper extremity robot on healthy adults. J Appl Biomech, 2009. 25(2): p. 103-10.
- 113. Vaisman, L., L. Dipietro, and H.I. Krebs, A comparative analysis of speed profile models for wrist pointing movements. IEEE Trans Neural Syst Rehabil Eng, 2013. 21(5): p. 756-66.
- Dipietro, L., A.M. Sabatini, and P. Dario, Evaluation of an instrumented glove for handmovement acquisition. J Rehabil Res Dev, 2003. 40(2): p. 179-89.



| HRP-503BIO | IMAS Optimization and Applicability in Acute and Subacute Stroke |
|---|---|

- 115. Sternad, D., et al., Transitions between discrete and rhythmic primitives in a unimanual task. Front Comput Neurosci, 2013. 7: p. 90.
- 116. Giacobbe, V., et al., Transcranial direct current stimulation (tDCS) and robotic practice in chronic stroke: the dimension of timing. NeuroRehabilitation, 2013. 33(1): p. 49-56.
- 117. Dipietro, L., et al. Effect of subthalamic nucleus stimulation on implicit motor learning. in Society for Neuroscience. 2012.
- 118. Krebs, H.I., et al., Autonomous Robots, 2003. 15(7): p. 7-20.
- 119. Finley, M.A., et al., Short-duration robotic therapy in stroke patients with severe upper-limb motor impairment. J Rehabil Res Dev, 2005. 42(5): p. 683-92.
- Dipietro, L., H. Poizner, and H.I. Krebs, Spatiotemporal dynamics of online motor correction processing revealed by high-density electroencephalography. J Cogn Neurosci, 2014. 26(9): p. 1966-80.
- 121. Dipietro, L., et al. Kinematic analysis of wrist motor learning. . in Society for Neuroscience. 2007.